CLINICAL TRIAL: NCT03245814
Title: Quantifying the Efficacy and Role of Service Dogs for Military Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Maggie O'Haire, Professor, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R21HD091896-01 (NIH); R21HD091896-01 (NIH)
Record Dates: First submitted 2017-07-05; First posted 2017-08-10 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: service dogs; human-animal interaction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Human-Animal Interaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinician Administered PTSD Scale for DSM-V (CAPS-5) assessments will be completed via telephone by a trained CAPS-5 rater who will be masked to the intervention and treatment arm of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Service Dog (Experimental): Participants in the service dog arm will receive unrestricted, non-study usual care, in addition to a trained service dog.
  Interventions: Behavioral: Service Dog
- Waitlist Control (No Intervention): Participants in the control arm will receive unrestricted, non-study usual care, while on the waitlist for a service dog.

INTERVENTIONS:
Behavioral: Service Dog — A service dog trained to perform tasks that are specific to PTSD
  Arms: Service Dog

SUMMARY:
The purpose of this study is to quantify the therapeutic efficacy and role of trained service dogs on socio-emotional functioning among military veterans with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
The long-term research goal is to evaluate the safety and efficacy of service dogs as a complementary intervention to enhance biopsychosocial functioning in special populations. The objective is to conduct a methodologically rigorous trial to quantify the therapeutic efficacy of service dogs on clinically-important outcomes for veterans with PTSD. Based on preliminary findings and qualitative reports, the central hypothesis is that military veterans with PTSD who are provided service dogs will experience reduced PTSD symptoms related to socio-emotional functioning and arousal modulation. The rationale for this research is that its successful completion will provide an evidence-based demonstration of the efficacy and role of an increasingly used yet poorly tested complementary intervention. The completion of this project is expected to established an initial demonstration of the therapeutic efficacy of service dogs in this population, as well as possible mechanisms of action via specific biological pathways and human-canine interaction profiles.

ELIGIBILITY:
Inclusion criteria for veterans into the study will include:

* Applied for and approved to receive a dog from K9s For Warriors
* Military service on or after September 11, 2001
* Honorable discharge or current honorable service
* Diagnosis of PTSD
* No conviction of any crimes against animals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite O'Haire, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leighton SC, Rodriguez KE, Jensen CL, MacLean EL, Davis LW, Ashbeck EL, Bedrick EJ, O'Haire ME. Service Dogs for Veterans and Military Members With Posttraumatic Stress Disorder: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2414686. doi: 10.1001/jamanetworkopen.2024.14686. PMID 38833250
- [Derived] Leighton SC, Rodriguez KE, Zhuang R, Jensen CL, Miller EA, Sabbaghi A, O'Haire ME. Psychiatric service dog placements are associated with better daily psychosocial functioning for military veterans with posttraumatic stress disorder. Psychol Trauma. 2024 Dec;16(Suppl 3):S707-S717. doi: 10.1037/tra0001543. Epub 2023 Jul 6. PMID 37410417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment, eligibility screening, and enrollment occurred between July 2017 and December 2019. Veterans were recruited through the database of an accredited nonprofit service dog organization, K9s For Warriors.
Pre-assignment Details: Of 200 participants recruited and screened, 170 met inclusion criteria and were enrolled and allocated.
Groups:
- Service Dog: Participants in the service dog arm received unrestricted, non-study usual care, in addition to a trained service dog.
  Service Dog: A service dog trained to perform tasks that are specific to PTSD
- Waitlist Control: Participants in the control arm received unrestricted, non-study usual care, while on the waitlist for a service dog.
Period: Overall Study
Arm/Group | Service Dog | Waitlist Control
Started | 91 | 79
Received Allocated Condition | 81 (Received service dog) | 75 (Remained on waiting list)
Completed | 76 | 67
Not Completed | 15 | 12
Not completed — Lost to Follow-up | 5 | 8
Not completed — Excluded (did not receive allocated condition) | 10 | 4

BASELINE CHARACTERISTICS:
Population: Based on a modified Intent-to-Treat analysis, in which participants were excluded if they did not receive the allocated condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Service Dog | Waitlist Control | Total
Number analyzed (Participants) | 81 | 75 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (8.2) | 38.2 (8.5) | 37.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 64 | 53 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 62 | 59 | 121
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 8 | 9 | 17
  White | 62 | 55 | 117
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 81 | 75 | 156
PTSD (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5); range 0-80; higher scores indicate worse outcome.
  units on a scale | 57.0 (11.3) | 55.7 (14.3) | 56.4 (12.8)
PTSD (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — Clinician-Administered PTSD Assessment for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition DSM-V (CAPS-5); range 0-80; higher scores indicate worse outcome.
  units on a scale | 42.0 (7.6) | 40.0 (7.0) | 41.1 (7.4)
Depression (PROMIS Depression) [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.0 - Emotional Distress - Depression 8a; T-score range 38 to 81; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
  T-score | 64.9 (7.8) | 62.7 (8.4) | 63.8 (8.1)
Anxiety (PROMIS Anxiety) [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.0 - Emotional Distress - Anxiety 8a; T-score range 37 to 83; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
  T-score | 68.2 (5.8) | 66.5 (5.5) | 67.4 (5.7)
PROMIS Social Isolation [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Social Isolation 8a; T-score range 33 to 76; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse outcome.
  T-score | 65.3 (8.2) | 62.7 (8.8) | 64.1 (8.6)
PROMIS Companionship [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Companionship 6a; T-score range 24 to 64; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better outcome
  T-score | 44.9 (10.7) | 46.9 (9.5) | 45.9 (10.1)
PROMIS Social Activities [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Ability to Participate in Social Roles and Activities 8a; T-score range 25 to 65; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better outcome.
  T-score | 50.8 (8.2) | 50.1 (6.3) | 50.5 (7.3)
VR-12 MCS [Mean (Standard Deviation); unit: units on a scale] — Veterans Rand 12-item Health Survey (VR-12) - Mental Health Component; range 0-100; higher scores indicate better outcome.
  units on a scale | 26.0 (11.3) | 28.2 (9.9) | 27.1 (10.7)
BSPW [Mean (Standard Deviation); unit: units on a scale] — Bradburn Scale of Psychological Wellbeing (BSPW); range -5 to 5; higher scores indicate better outcome.
  units on a scale | -2.7 (1.8) | -2.2 (1.9) | -2.4 (1.8)
SWLS [Mean (Standard Deviation); unit: units on a scale] — Satisfaction with Life Scale (SLS); range 3-35; higher scores indicate better outcome.
  units on a scale | 13.3 (6.3) | 13.8 (6.6) | 13.6 (6.4)
CD-RISC-10 [Mean (Standard Deviation); unit: units on a scale] — Connor-Davidson Resilience Scale (CDRS); range 0-40; higher scores indicate better outcome.
  units on a scale | 17.5 (7.5) | 20.8 (7.2) | 19.1 (7.5)
PROMIS Anger [Mean (Standard Deviation); unit: T-score] — Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.1 - Emotional Distress - Anger 5a; T-score range 32-82; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse outcome.
  T-score | 68.7 (9.1) | 64.9 (8.7) | 66.9 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Severity and Symptoms Via Self-report
Description: Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5); range 0-80; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | 41.9 (16.9) | 51.7 (16.1)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; Covariates included baseline score & demographic/clinical characteristics. Multiple imputation was used to account for uncertainty (missingness); Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.12 to 0.42]

2. Primary Outcome: PTSD Severity and Symptoms Via Clinician Rating
Description: Clinician-Administered PTSD Assessment for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition DSM-V (CAPS-5); range 0-80; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | 30.2 (10.2) | 36.9 (10.2)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; Covariates included baseline scores & demographic/clinical characteristics. Multiple imputation was used to account for uncertainty (missingness); Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.11 to 0.40]

3. Primary Outcome: Depression
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.0 - Emotional Distress - Depression 8a; T-score range 38 to 81; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Service Dog: Participants in the service dog arm will received, non-study usual care, in addition to a trained service dog.
  Service Dog: A service dog trained to perform tasks that are specific to PTSD
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 58.9 (9.5) | 61.4 (8.0)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = .02, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.23 to 0.86]

4. Primary Outcome: Anxiety
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.0 - Emotional Distress - Anxiety 8a; T-score range 37 to 83; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 62.1 (7.1) | 66.0 (5.4)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.13 to 0.50]

5. Secondary Outcome: Social Isolation
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Social Isolation 8a; T-score range 33 to 76; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 60.1 (10.8) | 62.8 (8.6)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.18 to 0.64]

6. Secondary Outcome: Companionship
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Companionship 6a; T-score range 24 to 64; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better outcome
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 48.5 (10.1) | 45.2 (9.3)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = .003, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [1.47 to 5.45]

7. Secondary Outcome: Ability to Participate in Social Activities
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v2.0 - Ability to Participate in Social Roles and Activities 8a; T-score range 25 to 65; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 45.2 (8.3) | 49.6 (6.3)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.12 to 0.48]

8. Secondary Outcome: Mental Health Quality of Life
Description: Veterans Rand 12-item Health Survey (VR-12) - Mental Health Component; range 0-100; higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | 36.3 (10.7) | 29.1 (10.4)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 3.84, 95% CI 2-sided [2.00 to 7.38]

9. Secondary Outcome: Psychological Well-being
Description: Bradburn Scale of Psychological Wellbeing (BSPW); range -5 to 5; higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | -0.6 (2.7) | -2.2 (2.2)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.49, 95% CI 2-sided [2.28 to 8.83]

10. Secondary Outcome: Life Satisfaction
Description: Satisfaction with Life Scale (SLS); range 3-35; higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | 19.7 (7.0) | 15.3 (6.9)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p < .001, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 3.73, 95% CI 2-sided [1.88 to 7.40]

11. Secondary Outcome: Resilience
Description: Connor-Davidson Resilience Scale (CDRS); range 0-40; higher scores indicate better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
units on a scale | 21.7 (6.3) | 20.8 (7.7)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = .02, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.22 to 4.47]

12. Secondary Outcome: Anger
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.1 - Emotional Distress - Anger 5a; T-score range 32-82; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 81 | 75
T-score | 61.2 (10.5) | 64.1 (10.0)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = .009, Ordinal cumulative probability model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.20 to 0.75]

13. Secondary Outcome: Daily Socio-emotional Experiences
Description: Ecological momentary assessment (EMA) Social interaction quality; range 0-6; higher score indicates better outcome.
Time Frame: 3 months
Population: This analysis was conducted with all participants who had available data based on initial group assignment. It differs from the other analyses in that it was done prior to the primary outcomes analysis and does not follow the same modified intent-to-treat analysis as conducted with the other outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Service Dog | Waitlist Control
Number analyzed (Participants) | 91 | 77
units on a scale | 4.2 (1.5) | 3.9 (1.5)
Statistical Analysis 1: Comparison: Service Dog vs Waitlist Control; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mixed effects regression models to account for repeated measures (multiple assessments per day) within individuals; Slope = 0.42, Standard Error of Mean 0.14

14. Other Pre Specified Outcome: Work and Activity Participation
Description: Work Productivity and Activity Impairment Questionnaire (WPAIQ)
Time Frame: 3 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Suicidal Ideation
Description: Columbia Suicide Severity Rating Scale (CSSRS)
Time Frame: 3 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Sleep Quality
Description: Pittsburgh Sleep Quality Assessment (PSQI)
Time Frame: 3 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Sleep Disturbance
Description: Patient Reported Outcome Measurement Information System (PROMIS) Adult Short Form (SF) v1.0 - Sleep Disturbance 8a
Time Frame: 3 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Sleep Actigraphy
Description: Actiwatch 2 (Philips Respironics)
Time Frame: 3 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Salivary Cortisol Awakening Response
Description: Passive drool method (Salimetrics)
Time Frame: 3 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Electrodermal Activity (Skin Conductance)
Description: Embrace wristband (Empatica, Inc.)
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected through passive surveillance. Participants spontaneously reported adverse events during study assessment periods (equivalent reporting opportunities across both groups) and during a 3-week on-site group class at the service dog organization (intervention group only).
Arm/Group | Service Dog | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/75
Serious Adverse Events (participants affected / at risk) | 4/81 | 6/75
Other Adverse Events (participants affected / at risk) | 1/81 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Service Dog (N=81) | Waitlist Control (N=75)
Inpatient hospitalization (Surgical and medical procedures) | 4 (4) | 6 (6) — Inpatient hospitalizations not related to the intervention or study (e.g., accidents, pre-existing condition treatment)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Service Dog (N=81) | Waitlist Control (N=75)
Dog bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03245814/Prot_SAP_000.pdf